CLINICAL TRIAL: NCT02784652
Title: Phase II Study of Efficacy of Radiotherapy in Combination With Zoledronic Acid on Pain Relief in Bone Metastasis Patients With Gastrointestinal Tumors
Brief Title: Efficacy of Radiotherapy in Combination With Zoledronic Acid in Bone Metastasis Patients With Gastrointestinal Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, Jinsil Seong, Professor in Dept. of Radiation Oncology, Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2014-0440; NCT02231476 (obsolete NCT alias)
Record Dates: First submitted 2016-05-01; First posted 2016-05-27 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Bone Metastasis; Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Zoledronic Acid; Radiotherapy

ARMS (1):
- RT & Zoledronic acid (Experimental): Radiotherapy: 5 days/ week, 3 Gy * 10-13 fractions or 4 Gy * 5 fractions, Zoleronic acid: every 4 weeks, 6 times, 4.0 mg iv
  Interventions: Drug: Zoledronic acid; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Zoledronic acid — Zoledronic acid: every 4 weeks, 6 times, 4.0 mg iv
  Other Names: Zolenic; Zometa
Radiation: Radiotherapy — Radiotherapy: 5 days/ week, 3 Gy * 10-13 fractions or 4 Gy * 5 fractions,

SUMMARY:
Bone metastasis causes bone destruction and skeletal related events (SRE) including compression fracture, hypercalcemia, and spinal cord compression. Therefore, palliative treatments for pain control and local control have become important and multidisciplinary multimodality approach is needed for treatment of bone metastasis.

The efficacy of radiotherapy (RT) for bone metastasis is well known. And the results that bisphosphonate decreases SRE in patients with solid tumor and multiple myeloma reported. In previous retrospective reports, the combination of local RT and systemic bisphosphonate was more effective than RT alone.

Therefore, Investigators designed a phase II study to evaluate the efficacy of RT in combination with zoledronic acid on pain relief and the safety of RT in bone metastasis patients with gastrointestinal tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with radiologic detectable bone metastasis (spine or non-spine)
* Patients with clinical diagnosis of gastrointestinal cancer: esophagus, stomach, colorectum, anus, liver, pancreas, gallbladder, biliary tract, etc.
* Patients over 20 years of age of both genders
* ECOG: 0 ~ 2
* Pain: worst pain score on BPI ≥3

Exclusion Criteria:

* Undetectable bone metastasis on radiologic study
* Patients who have previous surgery history at same site
* Patients who are considered surgery first: pathologic fracture, neurological or radiological evidence of spinal cord compression, impending pathologic fracture
* Patients who have hypersensitivity for zoledronic acid or other bisphosphonate
* Patients who have treatment history with zoledronic acid or other bisphosphonate
* Abnormal renal function or history of kidney transplantation
* Patients with metabolic bone disease
* Synchronous symptomatic brain metastasis
* Women who are pregnant, breast-feeding, or possible pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Pain relief rate | Change from baseline pain extent at 1,3,6 months

SECONDARY OUTCOMES:
skeletal related events (fracture and spinal cord compression) | at 18months after the IRB approval
  skeletal related events (SRE) (fracture, spinal cord compression due to metastasis requiring operation or radiotherapy. Occurence of pain is not regarded as SRE.) (SRE including fracture will be evaluated with plain X-ray at 1 month after completion of RT, and plain X-ray and MRI at 3 months after completion of RT.
  all imaging studies will be reviwed by clinician and radiologist.)
Overall survival | at 18months after the IRB approval

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, South Korea